CLINICAL TRIAL: NCT00001163
Title: Clinical, Laboratory, and Epidemiologic Characterization of Individuals and Families at High Risk of Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 780039; 78-C-0039; NCT00004007 (obsolete NCT alias)
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2026-01-05 (Actual); Status verified 2025-07-28

CONDITIONS: Hereditary Neoplasms; Cancer; Genetic Predisposition to Cancer; Environment
Keywords: Cancer; Genes/Genetics; Hereditary Neoplasms; Environment; Natural History
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: primary clinical; volunteers come from all U.S.

SUMMARY:
This is a clinical, epidemiologic, genetic, and laboratory study of individuals and families at high risk of cancer and selected tumors to investigate the genetic susceptibility and environmental exposures which may alter cancer risk. Families with multiple members who have an unusual pattern or number of cancers or tumors are evaluated clinically. This evaluation is specific for the type of cancer or tumor predominant in the family in order to determine the affection status of each individual for genetic epidemiologic studies. Genetic and environmental risk factor information specific for the tumor type is obtained.

Individuals with, or at high risk of, cancer because of their personal, familial, or environmental histories are identified by healthcare worker referral or by personal inquiry. Relevant etiologic risk factor information is documented through review of pathology specimens and medical, vital, and genealogical records. Selected individuals and family members are asked to complete questionnaires and to undergo clinical evaluations specific for the tumor of interest. They are also asked to donate biologic specimens to be used in the search for cancer etiology and mechanisms of carcinogenesis. No therapy beyond counseling and education for cancer prevention, risk reduction, and early detection will be given.

Genetic testing for tumor susceptibility gene(s) mutations and risk notification will be offered to study participants for whom a specific mutation predictive of disease has been identified in his/her family. This testing will only be offered when reasonable individual cancer risk estimates can be delivered, and only to those participants who choose to know their individual genetic status after appropriate education and counseling. The testing will be conducted exclusively in Clinical Laboratory Improvement Amendments (CLIA)-licensed laboratories. Genetic testing and risk notification are entirely optional and do not affect participation in other aspects of the protocol. A separate consent procedure and consent form will be used for genetic testing and risk notification related to these specific genes.

Once enrolled, study participants are monitored prospectively for the development of outcomes of interest, typically by means of periodic mail or telephone contact. In selected instances, subjects may return to the Clinical Center periodically for study-specific follow-up examinations. Although we do not offer specific anti-cancer therapy as part of this protocol, we provide assistance to insure that study participants who require treatment for tumor-related problems that develop during the course of the study are referred to appropriate healthcare providers. We remain available to study participants and their healthcare providers for advice and consultation related to the management of familial cancer/tumor predisposition.

DETAILED DESCRIPTION:
Background:

Persons may be prone to develop cancer for a variety of reasons including: inherited predisposition benign, premalignant, or malignant conditions; environmental exposures shared by family members; previous tumors, immune deficiency, or preneoplastic conditions.

Investigations of individuals and families at high risk of cancer often lead to etiologic clues that may be important in the sporadic counterparts of these cancers in the general population.

Identification of etiologically important genetic factors could inform chemoprevention trials, screening programs, and treatment of the studied cancer types.

Objectives:

To evaluate and define the clinical spectrum and natural history of disease in syndromes predisposing to cancer.

To evaluate potential precursor states of disease in families at risk.

To quantify risks of tumors in family members.

To map, clone, and determine function of tumor susceptibility genes.

To identify genetic determinants, environmental factors, and gene-environment interactions conferring cancer risk in individuals and families.

To evaluate gene-gene and gene-environment interactions in tumor formation.

To educate and counsel study participants about their tumor risk including prevention recommendations and early detection activities when known.

To develop educational materials for medical professionals and high-risk family members.

Eligibility:

Persons of any age will be considered for inclusion in the study because of either,

A family or personal medical history of neoplasia of an unusual type, pattern, or number; or,

Known or suspected factor(s) predisposing to neoplasia, either genetic and/or congenital factors, environmental exposure, or unusual demographic features.

Types of familial tumors that we are currently actively accruing include Cancers: bladder, bone, brain, chordoma, lung, nevoid basal cell carcinoma syndrome (NBCC).

Design:

This is a prospective study. Individuals and families are studied long-term, using a cohort approach.

The study design and clinical evaluation vary by the specific type of familial neoplasm being studied.

The overall approach to eligible study participants includes defining affection status, characterization of disease, localization of genetic loci, identification of genes, evaluation of phenotype/genotype correlations, estimation of risk of the disease associated with carrier status and identification of other risk factors that modify penetrance (genetic, environmental, host factors).

ELIGIBILITY:
* INCLUSION CRITERIA:

On referral, persons of any age will be considered for the inclusion in the study because of either:

A family or personal history of neoplasia of an unusual type, pattern, or number; OR,

known or suspected factor(s) predisposing to neoplasia, either genetic and/or congenital factors (birth defects, metabolic phenotype, chromosomal anomalies or Mendelian traits associated with tumors), environmental exposure (medications, occupation, radiation, diet, infectious agents, etc.), or unusual demographic features (very young age of onset, multiple tumors, etc.).

Personal and family medical history must be verified through questionnaires, interviews, and review of pathology slides and medical records. For familial neoplasms, two or more living affected cases among family members are required. The types of familial tumors that we are currently actively accruing include:

Familial Cancers: bladder, brain, chordoma, lung, nevoid basal cell carcinoma syndrome (NBCC)

Familial Benign Neoplasms: meningiomas, neurofibromatosis 2 (bilateral acoustic neurofibromatosis)

The types of familial tumors under active accrual and study are predominantly investigator-and hypothesis-driven. This approach permits GEB investigators to remain alert to the opportunities afforded by clusters of rare tumors in families and individuals, and to be more responsive to the dynamic research priorities in cancer genetics.

EXCLUSION CRITERIA:

Referred individuals and families for whom reported diagnoses cannot be verified.

Inability to provide informed consent.

Eligible for familial melanoma, lymphoproliferative, breast-ovarian cancer, or testicular cancer protocols.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary clinical; volunteers come from all U.S.
Sampling Method: Non-Probability Sample
Enrollment: 5201 (Actual)
Dates: Start 1985-04-02 (Actual)

PRIMARY OUTCOMES:
Defining the natural history of familial cancers and susceptibility states over multiple generations, identifying cancer susceptibility genes, and assessing gene-environment and gene-gene interactions | Ongoing
  New cancer development or current health status

CONTACTS AND LOCATIONS:
Overall Officials: Sharon A Savage, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Section 6.2 titled Data Sharing Plan in the protocol describes the plan for data sharing plans including human data sharing and genomic data sharing plan.@@@@@@Genotype and sequence data along with clinical phenotypes will be deposited in a genomic database in accordance with current NIH Genomic Data Sharing (GDS) Policy and the NIH Human Data Sharing Policy.@@@@@@The following human data generated in this research will be shared for future research as follows:@@@De-identified data in an NIH-funded or approved public repository.@@@@@@De-identified data in BTRIS (automatic for activities in the Clinical Center)@@@@@@De-identified or identified data with approved outside collaborators under appropriate agreements.@@@@@@The data will be shared at the time of publication or shortly after.@@@@@@Unlinked genomic data will be deposited in public genomic databases such as dbGaP in compliance with the NIH Genomic Data Sharing Policy.
Supporting Information: SAP, ICF
Time Frame: The data will be shared at the time of publication or shortly after.
Access Criteria: Section 6.2 titled Data Sharing Plan in the protocol describes the plan for data sharing plans including human data sharing and genomic data sharing plan.

REFERENCES:
- [Background] Pathak A, Seipel K, Pemov A, Dewan R, Brown C, Ravichandran S, Luke BT, Malasky M, Suman S, Yeager M; NCI DCEG Cancer Genomics Research Laboratory; NCI DCEG Cancer Sequencing Working Group; Gatti RA, Caporaso NE, Mulvihill JJ, Goldin LR, Pabst T, McMaster ML, Stewart DR. Whole exome sequencing reveals a C-terminal germline variant in CEBPA-associated acute myeloid leukemia: 45-year follow up of a large family. Haematologica. 2016 Jul;101(7):846-52. doi: 10.3324/haematol.2015.130799. Epub 2015 Dec 31. PMID 26721895
- [Background] Pathak A, Pemov A, McMaster ML, Dewan R, Ravichandran S, Pak E, Dutra A, Lee HJ, Vogt A, Zhang X, Yeager M, Anderson S, Kirby M; NCI DCEG Cancer Genomics Research Laboratory; NCI DCEG Cancer Sequencing Working Group; Caporaso N, Greene MH, Goldin LR, Stewart DR. Juvenile myelomonocytic leukemia due to a germline CBL Y371C mutation: 35-year follow-up of a large family. Hum Genet. 2015 Jul;134(7):775-87. doi: 10.1007/s00439-015-1550-9. Epub 2015 May 5. PMID 25939664
- [Derived] Korde LA, Mueller CM, Loud JT, Struewing JP, Nichols K, Greene MH, Mai PL. No evidence of excess breast cancer risk among mutation-negative women from BRCA mutation-positive families. Breast Cancer Res Treat. 2011 Jan;125(1):169-73. doi: 10.1007/s10549-010-0923-y. Epub 2010 May 11. PMID 20458532
- [Derived] Koehly LM, Peters JA, Kenen R, Hoskins LM, Ersig AL, Kuhn NR, Loud JT, Greene MH. Characteristics of health information gatherers, disseminators, and blockers within families at risk of hereditary cancer: implications for family health communication interventions. Am J Public Health. 2009 Dec;99(12):2203-9. doi: 10.2105/AJPH.2008.154096. Epub 2009 Oct 15. PMID 19833996
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_1978-C-0039.html